CLINICAL TRIAL: NCT05685602
Title: A Phase I Clinical Trial of CA-4948 in Combination With Gemcitabine and Nab-Paclitaxel in Metastatic or Unresectable Pancreatic Ductal Carcinoma
Brief Title: CA-4948 Added to Standard Chemotherapy to Treat Metastatic or Unresectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-08984; NCI-2022-08984 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 202304010; 10522 (Other: Yale University Cancer Center LAO); 10522 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2023-01-13; First posted 2023-01-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; Specimen Handling; CA-4948; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CA-4948, gemcitabine, nab-paclitaxel) (Experimental): Patients receive CA-4948 PO BID on days 1-21 or 1-28 of each cycle, gemcitabine IV over 30-60 minutes on days 1 and 8 or 1, 8, and 15 of each cycle, and nab-paclitaxel IV over 30-40 minutes on days 1 and 8 or 1, 8, and 15 of each cycle. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, tumor biopsies, and blood sample collection throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Emavusertib; Drug: Gemcitabine Hydrochloride; Drug: Nab-paclitaxel

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Emavusertib — Given PO
  Other Names: AU 4948; AU-4948; CA 4948; CA-4948; CA4948; Interleukin-1 Receptor-associated Kinase 4 Inhibitor CA-4948; IRAK4 Inhibitor CA-4948
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of emavusertib (CA-4948) in combination with gemcitabine and nab-paclitaxel in treating patients with pancreatic ductal adenocarcinoma that has spread from where it first started (primary site) to other places in the body (metastatic) or cannot be removed by surgery (unresectable). CA-4948 is in a class of medications called kinase inhibitors. It works by blocking the action of abnormal proteins called interleukin-1 receptor-associated kinase 4 (IRAK4) and FMS-like tyrosine kinase 3 (FLT3) that signal cells to multiply. This may help keep cancer cells from growing. The usual approach for patients with pancreatic ductal adenocarcinoma is treatment with chemotherapy drugs gemcitabine and nab-paclitaxel. Gemcitabine is a chemotherapy drug that blocks the cells from making DNA and may kill cancer cells. Paclitaxel is in a class of medications called anti-microtubule agents. It stops cancer cells from growing and dividing and may kill them. Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of paclitaxel which may have fewer side effects and work better than other forms of paclitaxel. Giving CA-4948 in combination with gemcitabine and nab-paclitaxel may shrink or stabilize metastatic or unresectable pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess dose limiting toxicities and determine the recommended phase 2 dose of emavusertib (CA--4948) in combination with chemotherapy in patients with pancreatic ductal adenocarcinoma.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the safety and tolerability of the combination of CA-4948 and chemotherapy.

III. To determine preliminary signals of efficacy, as measured by objective response rate (ORR), CA-4948 response, progression free survival (PFS), and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To evaluate pharmacodynamic effect of CA-4948 in combination with chemotherapy.

II. To evaluate pharmacokinetics of CA-4948 in combination with chemotherapy. III. To explore biomarkers and genomic alterations associated with treatment response.

OUTLINE: This is a dose-escalation study of CA-4948 in combination with fixed-dose gemcitabine and nab-paclitaxel followed by a dose-expansion study.

Patients receive CA-4948 orally (PO) twice daily (BID) on days 1-21 or 1-28 of each cycle, gemcitabine intravenously (IV) over 30-60 minutes on days 1 and 8 or 1, 8, and 15 of each cycle, and nab-paclitaxel IV over 30-40 minutes on days 1 and 8 or 1, 8, and 15 of each cycle. Cycles repeat every 21 or 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), tumor biopsies, and blood sample collection throughout the trial.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the pancreas that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have had disease progression on or after fluorouracil (5-FU)-based therapy for metastatic or unresectable pancreatic ductal adenocarcinoma (PDAC). If received gemcitabine-based regimen as adjuvant therapy, then gemcitabine and nab-paclitaxel (if used) should be >12 months from study enrollment. Prior use of gemcitabine/nab-paclitaxel for metastatic or unresectable disease is not allowed
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of CA-4948 in combination with gemcitabine and nab-paclitaxel in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 60 mL/min (based on the calculated Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] glomerular filtration rate estimation)
* Creatine phosphokinase (CPK) elevation at the screening < grade 2 (creatine phosphokinase [CPK] =< 2.5 ULN)
* Patients on a cholesterol lowering statin must be on a stable dose with no dose changes within 3 weeks prior to study start
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial as long as their anti-retroviral therapy does not have the potential for drug-drug interactions as judged by the treating investigator
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after at least 4 weeks following central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have lesions amenable to research biopsy for those enrolling to the expansion cohort. The biopsy should be deemed feasible and safe for pre-biopsy lesion assessment criteria
* The effects of CA-4948, nab-paclitaxel, and gemcitabine on the developing human fetus are unknown. For this reason and because gemcitabine is known to be teratogenic, embryotoxic, and fetotoxic in mice and rabbits, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 90 days after completion of CA-4948, nab-paclitaxel, and gemcitabine administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of CA-4948, nab-paclitaxel, and gemcitabine administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible
* Patients must have measurable disease per Response Evaluable Criteria in Solid Tumors (RECIST) 1.1

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from clinically significant adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of neuropathy, which should resolve to grade 2, or alopecia
* History of other malignancy with the exception of 1) malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease; 2) or known indolent malignancies that do not require treatment and will likely not alter the course of treatment of disease under treatment
* History of allogeneic organ or stem cell transplant
* Current use or anticipated need for alternative, holistic, naturopathic, or botanical formulations used for the purpose of cancer treatment
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CA-4948 or other agents used in study
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible due to CA-4948 and nab-paclitaxel. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because gemcitabine is nucleoside analogue with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with gemcitabine, breastfeeding should be discontinued if the mother is treated with gemcitabine. These potential risks may also apply to other agents used in this study
* Prolonged Fridericia's correction formula (QTcF) (> 470 in females, > 450 in males) on screening electrocardiogram (ECG)
* Gastrointestinal condition which could impair absorption of CA-4948 or inability to ingest CA-4948
* Severe obstructive pulmonary disease or interstitial lung disease
* History of rhabdomyolysis or elevated creatine phosphokinase (CPK)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rate | Up to 1 year
  Done to determine the maximum tolerated dose for the combination of CA-4948 and gemcitabine/nab-paclitaxel chemotherapy backbone. Data analysis of the study will be descriptive in nature. Demographic and clinical characteristics of the sample, toxicity by severity, as well as loss to follow-up will be summarized using descriptive statistics. Safety endpoints will be listed for each dose level.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 1 year
  Tabulations of adverse events will be produced by severity and by relationship to study drug.
Overall response rate (ORR) | Up to 1 year
  For efficacy data in the expansion cohort, ORR and its 95% confidence interval will be calculated.
Progression-free survival (PFS) | From start of study treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  Will be described using Kaplan-Meier product limit methods.
Overall survival (OS) | Up to 1 year
  Will be described using Kaplan-Meier product limit methods.

OTHER OUTCOMES:
Pharmacodynamic effect of CA-4948 in combination with chemotherapy | Up to 1 year
  Pharmacodynamic indices from biopsies obtained from expansion cohorts will be summarized using descriptive statistics (means, median, and standard deviations) at each measurement time point and the change will be compared by paired t-test or Wilcoxon rank-sum test as appropriate.
Pharmacokinetics (PK) of both CA-4948 and nab-paclitaxel | Cycle 1 day 1 (C1D1) (pre-dose, 0.5, 1, 2, 4, 6, 8 hours [h]), C1D8 (pre-dose), C2D1 (pre-dose, 0.5, 1, 2, 4, 6, 8h), C2D2: (24h post C2D1 dose), C2D8 (pre-dose), C3D1 (pre-dose), C3D17 (+/- 3 d)
  Done to confirm whether a clinically relevant drug-drug interaction occurs. Plasma concentration-time curves will be analyzed by noncompartmental methods using routines supplied in the Phoenix WinNonlin Professional software package. Exposure obtained by noncompartmental methods will also be compared to toxicity and efficacy outcomes using graphical and statistical programs. A formal population PK or exposure-response analyses may be conducted based on these initial findings.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Grierson, Principal Investigator — Yale University Cancer Center LAO
Locations (26):
- United States (26):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm